CLINICAL TRIAL: NCT01619657
Title: Randomized, Double-blind, Controlled Pilot Study on Safety of Hypertonic Saline as Preventive Inhalation Therapy in Newborns and Infants With Cystic Fibrosis
Brief Title: Preventive Inhalation of Hypertonic Saline in Infants With Cystic Fibrosis
Acronym: PRESIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Center for Lung Research (Other)
Responsible Party: Principal Investigator, Marcus A. Mall, MD, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UKH-PIHSNC-1
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Cystic Fibrosis Lung Disease
Keywords: Cystic Fibrosis; Hypertonic Saline; Infant; Newborn; Prevention
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypertonic Saline (Experimental): Inhalation with 6% Hypertonic Saline twice daily over 1 year
  Interventions: Drug: 6% Hypertonic Saline (HS), 4mL
- Isotonic Saline (Active Comparator): Inhalation with 0.9% Isotonic Saline twice daily over 1 year
  Interventions: Drug: 0.9% Isotonic Saline (IS), 4mL

INTERVENTIONS:
Drug: 6% Hypertonic Saline (HS), 4mL — Administered via inhalation twice daily for 52 weeks. The delivery system is a PARI LC SPRINT® Junior nebulizer with a baby bend, size-adapted PARI® Baby face mask size 0-3, connection tubing (2.2m) and a PARI JuniorBOY® SX compressor.
  Other Names: MucoClear® 6%
  Arms: Hypertonic Saline
Drug: 0.9% Isotonic Saline (IS), 4mL — Administered via inhalation twice daily for 52 weeks. The delivery system is a PARI LC SPRINT® Junior nebulizer with a baby bend, size-adapted PARI® Baby face mask size 0-3, connection tubing (2.2m) and a PARI JuniorBOY® SX compressor.
  Other Names: Normal Saline
  Arms: Isotonic Saline

SUMMARY:
The purpose of this study is to assess whether 6% hypertonic saline (HS) is a safe and effective preventive therapy in newborns and infants with cystic fibrosis (CF).

DETAILED DESCRIPTION:
Cystic fibrosis (CF) remains one of the most common lethal genetic diseases in Europe and North America. Despite a substantial increase in life expectancy over the past decades, many CF patients still die during young adulthood due to chronic progressive CF lung disease that is caused by defective fluid transport by airway epithelia causing dehydration of airway surfaces, which in turn leads to impaired mucociliary clearance, chronic airway mucus obstruction, inflammation and infection. Recent evidence from studies in a mouse model of CF lung disease suggest that preventive improvement of airway surface hydration may be an effective treatment of early and reversible mucus obstruction and inflammation, and thus delay or ameliorate progressive damage in lungs of CF patients. Hypertonic saline (HS) is an osmotic agent that improves airway surface hydration, and inhalation of 6% HS is already an established, safe, and effective maintenance therapy that improves mucociliary clearance and lung function, and reduces pulmonary exacerbations in older children (> 6 years) and adults with chronic CF lung disease and fixed lung damage. However, the effect of HS as a preventive therapy has not been studied, and no other therapies are available for preventive improvement of airway dehydration and mucociliary dysfunction in CF.

This investigator initiated clinical trial is a monocentric, randomized, double-blind, controlled pilot study on safety and efficacy of a preventive and early inhalation with HS in newborns and infants with CF who are diagnosed in the newborn period either by CF newborn screening (CF-NBS) or for another reason (e.g. meconium ileus) and are younger than 4 months of age at the time of enrolment. Participating patients will be randomized to 6% HS or 0.9% isotonic saline (IS) as active comparator. In both groups, patients will inhale their study solution twice daily over 52 weeks. At the beginning, during and at the end of the study, different measurements will be undertaken to determine effects of HS on safety, radiologic and/or functional alterations of the lung, number of exacerbations, time to first detection of a CF pathogen, and health-related quality of life. We expect that the results of this study will provide first evidence on the safety and efficacy of a preventive therapy that improves airway surface hydration and targets a CF basic defect and may thus delay and/or ameliorate chronic damage of the lungs of patients with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CF established in neonatal period either via CF newborn screening (NBS) or because of symptoms typical for CF (e.g. meconium ileus), positive family history or positive prenatal screening and fulfilling at least one of the following three criteria:

   * sweat chloride ≥ 60mEq/L
   * two CF causing mutations of CFTR gen
   * alterations of transepithelial potential difference of nasal or rectal epithelia typical for CF.
2. Age at enrolment is 0 to 4 months.
3. Patient's and parent's ability to comply with medication use, study visits, and study procedures is judged by the investigator (therefore parents have to understand the character of the study and individual consequences).
4. Participation in this study is voluntary. Only patients, whose parents or legal guardians gave written consent, are included.

Exclusion Criteria:

1. Born < 30 weeks gestation.
2. Prolonged mechanical ventilation in the first 3 months of life.
3. A significant medical disease or condition other than CF likely to interfere with the child's ability to complete the entire protocol.
4. Previous major surgery except for meconium ileus.
5. Other major organ dysfunction, excluding pancreatic or hepatic dysfunction or another condition due to cystic fibrosis.
6. Physical findings that would compromise the safety of the subject or the quality of the study data as determined by investigator.
7. History of adverse reaction to sedation.
8. Known hypersensitivity to study treatment.
9. Participation in other interventional studies at the same time.

Criteria, which lead to a displacement of the procedures in sedation until the child has recovered:

* Clinically significant upper airway obstruction as determined by investigator (e.g. severe laryngomalacia, markedly enlarged tonsils, significant snoring, diagnosed obstructive sleep apnoea).
* Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate with onset in 2 weeks preceding visit.
* Oxygen saturation <95% before initial pulmonary function test or initial MRI.
* Severe gastroesophageal reflux, defined as persistent frequent emesis despite anti-reflux therapy.

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2012-06; Primary Completion 2016-11 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of patients in both treatment groups with adverse events (AEs) and serious adverse events (SAEs) | during the 52 week treatment period
  Safety of inhalation with HS and IS in newborns and infants with CF assessed by proportion of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Rate of protocol-defined pulmonary exacerbations | during the 52 week treatment period
  Rate of protocol-defined pulmonary exacerbations requiring treatment with oral, inhaled or intravenous antibiotics between subjects randomized to HS and IS
Time to first pulmonary exacerbation in both treatment groups | during the 52 week treatment period
Proportion of children with morphological and/or functional changes due to CF lung disease at baseline and after 1 year of inhalation | during the 52 week treatment period
  Proportion of children with morphological and/or functional changes due to CF lung disease at baseline and after 1 year of inhalation according to magnetic resonance imaging (MRI) chest score and chest x-ray (CXR) Chrispin-Norman score in both groups (HS vs. IS)
Extent and severity of bronchial dilatation | during the 52 week treatment period
  Extent and severity of bronchial dilatation after MRI and CXR scores at baseline and after 1 year of inhalation in both groups
Proportion of children with impairments in lung function | during the 52 week treatment period
  Proportion of children with impairments in lung function determined via multiple breath washout at baseline, after 3, 6, 9, and 12 months of inhalation in both groups
Severity of impairment in lung function test | during the 52 week treatment period
  Severity of impairment in lung function test at baseline, after 3, 6, 9, and 12 months of inhalation in both groups
Health-related quality of life | during the 52 week treatment period
  Health-related quality of life as assessed by scores from Cystic Fibrosis Questionnaire - Revised Parent Report (CFQ-R, German version), administered quarterly
Change in anthropometric and basic respiratory parameters | during the 52 week treatment period
  Change in weight, height, body mass-index, weight-for-height, resting respiratory rate, and room air oxygen saturation
Proportion of patients with new isolation of CF pathogen | during the 52 week treatment period
  Among participants from whom Pseudomonas aeruginosa or other CF pathogens were not isolated from respiratory cultures prior to enrolment, the proportion from whom these organisms are isolated from clinically collected respiratory cultures
Time to first isolation of a CF pathogen | during the 52 week treatment period
  Time to acquisition of a CF pathogen is going to be compared between both treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Marcus A Mall, MD, Principal Investigator — University Hospital Heidelberg
Locations (4):
- Germany (4):
  - University Children's Hospital Heidelberg, Cystic Fibrosis Centre, Heidelberg, Baden-Wurttemberg
  - University Hospital Gießen and Marburg GmbH, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - University Children's Hospital Schleswig-Holstein, Lübeck

REFERENCES:
- [Derived] Wark P, McDonald VM, Smith S. Nebulised hypertonic saline for cystic fibrosis. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD001506. doi: 10.1002/14651858.CD001506.pub5. PMID 37319354
- [Derived] Stahl M, Wielputz MO, Ricklefs I, Dopfer C, Barth S, Schlegtendal A, Graeber SY, Sommerburg O, Diekmann G, Husing J, Koerner-Rettberg C, Nahrlich L, Dittrich AM, Kopp MV, Mall MA. Preventive Inhalation of Hypertonic Saline in Infants with Cystic Fibrosis (PRESIS). A Randomized, Double-Blind, Controlled Study. Am J Respir Crit Care Med. 2019 May 15;199(10):1238-1248. doi: 10.1164/rccm.201807-1203OC. PMID 30409023